CLINICAL TRIAL: NCT07309146
Title: Evaluation of the Quantity and Quality of Human Breast Milk Collected in a Single-center Milk Bank Over the Last Five Years
Brief Title: Single-center Evaluation of Human Milk Quantity and Quality Over Five Years
Acronym: HUMBLE
Status: Not yet recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Nemocnice České Budějovice, České Budějovice, Czechia (Unknown)
Responsible Party: Principal Investigator, Marek Petras, Principal Investigator, Charles University, Czech Republic
Other Study IDs: HUMBLE
Record Dates: First submitted 2025-12-04; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Lactating Women - Human Milk Donors
Keywords: donor human milk; human milk bank; milk donation; milk volume; milk quality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Human Milk Donors: Lactating women who donated human milk to the hospital-based human milk bank at České Budějovice Hospital between 2021 and 2025.
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — Retrospective observational study based on routinely collected clinical and milk bank data; no experimental procedure, treatment, or behavioral intervention is administered.

SUMMARY:
This single-center retrospective observational study includes all human milk donors collaborating with the milk bank at České Budějovice Hospital between 2021 and 2025. Using anonymized data extracted from the hospital database, the study will quantify the frequency of donations and the individual and cumulative volume of donated human milk and will assess the impact of key maternal and perinatal factors - including age, BMI, parity, mode of delivery, and timing of donations - on the quantity and quality of donated milk, based on routine biochemical and microbiological parameters.

DETAILED DESCRIPTION:
Donor human milk is a key component of nutritional care for preterm and high-risk neonates when mother's own milk is unavailable or insufficient. A better under-standing of which factors are associated with higher or lower donated volumes, and with favorable biochemical and microbiological milk characteristics, may help optimize several aspects of milk bank practice. This study aims to characterize a five-year experience from a single hospital-based human milk bank in terms of donation pat-terns and donated milk volume. It also aims to evaluate the relationship between key maternal and perinatal characteristics and both the quantity and routinely assessed quality of donated human milk.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women who donated human milk to the hospital-based human milk bank at České Budějovice Hospital during the period 2021-2025.
* Accepted as donors according to local eligibility criteria for human milk donation.
* At least one recorded donation of human milk with available data on donation date and volume in the milk bank database.
* Availability of basic maternal and perinatal data (e.g., age, BMI, parity, mode of delivery, timing of donation) in the hospital information sys-tem.

Exclusion Criteria:

* Donors with no recorded volume or date of human milk donation in the milk bank database.
* Records with evident data errors or inconsistencies that cannot be reliably corrected (e.g., implausible dates or volumes).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Lactating women who donated human milk to the hospital-based human milk bank at České Budějovice Hospital between 2021 and 2025. All donors met the local eligi-bility criteria for milk donation and collaborated with the milk bank during the de-fined period.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Donation intensity | Assessed at the end of each donor's donation period (from first to last recorded donation), within January 1, 2021 to December 31, 2025.
  Donation intensity, defined as the cumulative volume of donated human milk per donor (mL) and the number of donation episodes per donor over the individual donation period within the 5-year study window (2021-2025).

SECONDARY OUTCOMES:
Quality of donated human milk | Assessed at the end of each donor's donation period (from first to last recorded donation), within January 1, 2021 to December 31, 2025.
  Quality of donated human milk, assessed by routine biochemical composition parameters and microbiological safety indicators over the individual donation period within the 5-year study window (2021-2025). Biochemical composition parameters: fat (g/L), protein (g/L), carbohydrate (g/L), and calculated energy content (kcal/100 mL) Microbiological safety indicators: total viable bacterial count (CFU/mL) and culture result classified as pass/fail according to the milk bank's routine acceptance criteria

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Dlouhý, PhD, Study Director — Third Faculty of Medicine, Charles University, Prague, Czech Republic
Locations (1):
- Department of Epidemiology and Biostatistics, Third Faculty of Medicine, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of donor information, absence of explicit consent for external data sharing, and restrictions imposed by local regulations and GDPR.